CLINICAL TRIAL: NCT00365820
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Phase II/III Study to Evaluate the Efficacy and Safety of Tegaserod and Placebo Given Orally for 12 Weeks for the Treatment of Opioid-induced Constipation (OIC) in Patients With Chronic Non-cancer Pain
Brief Title: Efficacy and Safety of Tegaserod in Opioid-induced Constipation in Patients With Non-cancer Pain
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This study was terminated early as a result of regulatory action suspending tegaserod use in 2007
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919N2201
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Constipation
Keywords: Opioid, constipation, tegaserod; Opioid-induced constipation
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study will evaluate the efficacy and safety of tegaserod in opioid-induced constipation in patients with non-cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients 18 years of age or older.
2. Patients with chronic non-cancer pain that necessitates the use of non-injectable opioid analgesics. The equivalent dose of 300 mg morphine per day is the maximum opioid analgesic dose allowed. In general, patients should be using opioids on a daily basis.
3. Chronic pain which has been present for a minimum of 3 months which needs the chronic use of opioids for pain relief.
4. Constipation, according to the investigator's clinical judgment, that is resulting from opioid use for non-cancer chronic pain. Opioid-induced constipation (OIC) is defined as follows:

   * less than 3 spontaneous bowel movements per week and at least one of the following on at least 25% of occasions:

     1. hard or very hard stools
     2. sensation of incomplete evacuation
     3. straining while having a bowel movement

Exclusion Criteria:

1. Patients who are receiving opioids for abdominal pain or connective tissue disorders.
2. Planned discontinuation or an increase or decrease by more than 30% of the current opioid dose
3. Patients who underwent major surgery within 3 months prior to screening.
4. Patients with a history of prior chronic constipation (CC) that was present for more than three months and that was not related to opioid use.
5. Patients with a current diagnosis of irritable bowel syndrome (IBS) constipation predominant or alternators.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 670
Dates: Start 2006-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of bowel movements over weeks 1-4

SECONDARY OUTCOMES:
Change from baseline in the number of bowel movements over weeks 1-12
Change from baseline in abdominal distension/bloating over weeks 1-12
Change from baseline in abdominal discomfort/pain over weeks 1-12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (55):
- United States (55):
  - Investigative Site, Mobile, Alabama
  - Investigative Site, Phoenix, Arizona
  - Investigative Site, Tucson, Arizona
  - Investigative Site, North Little Rock, Arkansas
  - Investigative Site, Buena Park, California
  - Investigative Site, Downey, California
  - Investigative Site, Encinitas, California
  - Investigative Site, Fountain Valley, California
  - Investigative Site, La Jolla, California
  - Investigative Site, Los Angeles, California
  - Investigative Site, Mission Viejo, California
  - Investigative Site, San Diego, California
  - Investigative Site, San Francisco, California
  - Investigative Site, Torrance, California
  - Investigative Site, Northglenn, Colorado
  - Investigative Site, Bristol, Connecticut
  - Investigative Site, DeLand, Florida
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Largo, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, New Smyrna Beach, Florida
  - Investigative Site, Springhill, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Belleville, Illinois
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Avon, Indiana
  - Investigative Site, Evansville, Indiana
  - Investigative Site, Indianapolis, Indiana
  - Investigative Site, Overland Park, Kansas
  - Investigative Site, Prairie Village, Kansas
  - Investigative Site, Shreveport, Louisiana
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Omaha, Nebraska
  - Investigative Site, Pahrump, Nevada
  - Novartis Pharmaceutical Corporation, East Hanover, New Jersey
  - Investigative Site, New York, New York
  - Investigative Site, North Massapequa, New York
  - Investigative Site, Charlotte, North Carolina
  - Investigative Site, Greensboro, North Carolina
  - Investigative Site, Monroe, North Carolina
  - Investigative Site, Winston-Salem, North Carolina
  - Investigative Site, Dayton, Ohio
  - Investigative Site, Oklahoma City, Oklahoma
  - Investigative Site, Portland, Oregon
  - Investigative Site, Hershey, Pennsylvania
  - Investigative Site, Levittown, Pennsylvania
  - Investigative Site, Chattanooga, Tennessee
  - Investigative Site, Beaumont, Texas
  - Investigative Site, Colleyville, Texas
  - Investigative Site, Corsicana, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, San Antonio, Texas
  - Investigative Site, Salt Lake City, Utah
  - Investigative Site, Charlottesville, Virginia
  - Investigative Site, Seattle, Washington